CLINICAL TRIAL: NCT04450992
Title: TRACK-MSA: An Observational Longitudinal Oligo-Center Study to Define Clinical, Biofluid, Imaging and Digital Outcome Measures in Multiple System Atrophy
Brief Title: TRACK-MSA: A Longitudinal Study to Define Outcome Measures in Multiple System Atrophy
Status: Completed | Type: Observational
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Other Study IDs: S19-01846
Record Dates: First submitted 2020-06-25; First posted 2020-06-30 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Multiple System Atrophy
MeSH Terms: conditions — Multiple System Atrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biomarker analysis will be focused on measuring the levels of neurofilament light chain (NfL) in serum and/or plasma, which is one of the most promising blood biomarkers in MSA.
  Analysis of CSF may include but is not limited to the following biomarkers: total alpha synuclein, aggregated alpha synuclein Tau/phosphorylated Tau, neurofilament light chain, neurofilament heavy chain, and catecholamines (dopamine, norepinephrine, DOPAC, DHPG).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
TRACK-MSA is an observational, non-interventional, longitudinal natural history study to define changes in clinical, neurological, blood, CSF, and neuroimaging biomarkers in patients with multiple system atrophy (MSA) comparing baseline to 6-month and 1-year assessments. The study will enroll 50 patients with MSA-P or MSA-C at 2 or more participating sites.

DETAILED DESCRIPTION:
TRACK-MSA is designed to relate phenotypic characteristics of participants with MSA using several modalities (i.e., clinical, quantitative motor, imaging, laboratory) in order to relate phenotypic characteristics with data derived from the study of blood and CSF ("wet biomarkers") and imaging or wearables ("dry biomarkers").

It is possible that the cohort enrolled in this study will, after study completion, be recruited into the earliest multicenter biomarker-driven clinical trials of disease modifying agents for MSA. As such, the data collected in the TRACK-MSA study could constitute a valuable observational non-interventional arm of potential disease-modifying treatments.

The objective of the study will therefore be to determine the combination of measures that most sensitively detects changes over the natural course of MSA, with a goal of validating these measures for use in future clinical trials.

TRACK-MSA will be a 1-year observational, longitudinal, non-interventional natural history study of patients with MSA. The study will be carried out at least at 2 sites (NYU being the primary site). All participants will be assessed at baseline, 6-month and 1-year visits. Participants will undergo clinical, neurological, quantitative motor, MRI assessments, in addition to donating blood and CSF samples at some or all of the visits.

For a given participant, the same investigator should carry out the clinical assessment throughout the study where possible.

It is anticipated that the study will complete enrollment in 2 years since startup, and complete all the follow-up evaluations within 3 years from startup.

ELIGIBILITY:
Inclusion Criteria:

- 1. Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use confidential health information in accordance with applicable privacy regulations 2. Diagnosis of probable or possible multiple system atrophy (MSA-P or MSA-C) according to current consensus diagnostic criteria [8].

3. Aged 40-80 with anticipated survival of at least 3 years (in the opinion of the Investigator) 4. Able to walk for, at least, 10 meters with or without assistance 5. Willingness and ability to participate in all study procedures. 6. Ability to tolerate and no contraindications for brain MRI. 7. Ability to tolerate and no contraindications for CSF collection. Participants with contraindication to the CSF procedure will be given the option to participate in the study and opt out the CSF collection. An effort will be made to ensure that at least 50% of patients enrolled in the study undergo CSF collection.

Exclusion Criteria:

* 1. Presence of supranuclear gaze palsy. 2. Known presence of hyposmia (i.e., reduced ability to smell and detect odors).

  3. Presence of cognitive dysfunction (defined as MoCA score <20). 4. Severe-to-complete dependence on caregivers (score >3 on UMSARS Part IV, Global Disability), severe impairment of swallowing (score ≥3 on UMSARS Part I, Question 2), or frequent falls (score ≥3 on UMSARS Part I, Question 8) at Baseline.

  5. Family history or a known genetic cause of ataxia or parkinsonism. 6. Clinically significant neuropathy. 7. Hallucinations not induced by drugs. 8. Unstable psychiatric illness, including psychosis, suicidal ideation, or untreated major depression within 90 days before Baseline, as determined by the Investigator.

  9. History or Baseline MRI results showing evidence of structural abnormalities that could contribute to the participant's clinical state other than findings typical of MSA, or any finding that might pose a risk to the participant.

  10. Any contraindications to having a brain MRI (e.g., pacemaker; MRI-incompatible aneurysm clips, artificial heart valves, or other metal foreign body; claustrophobia that cannot be medically managed without requiring general anesthesia, etc.).

  11. Transient ischemic attack or stroke, or any unexplained loss of consciousness within 1 year before Baseline.

  12. History of any brain surgery for MSA (e.g., pallidotomy, deep brain stimulation, or fetal tissue transplant) or a history of focused ultrasound treatment or neuromodulation procedures, including but not limited to transcranial magnetic stimulation (TMS) and transcranial direct or alternating current stimulation (tDCS/tACS) that have been performed within 90 days of Baseline.

Infection Risk 13. History of human immunodeficiency virus or hepatitis C virus antibody. 14. Chronic, recurrent, or serious infection (e.g., pneumonia, septicemia, recurrent urinary tract infection), as determined by the Investigator, within 8 weeks before Day 1.

Cardiovascular 15. History of unstable angina, myocardial infarction, chronic heart failure (New York Heart Association Class 3 or 4), or clinically significant conduction abnormalities (e.g., unstable atrial fibrillation) within 1 year before Baseline.

16. Chronic, sustained, uncontrolled supine hypertension (unrelated to pharmacological treatment of orthostatic hypotension) defined by an average of three SBP readings of >180 mmHg or DBP readings of >110 mmHg at baseline.

17. In participants treated pharmacologically for orthostatic hypotension, any documented sitting or standing SBP reading ≥180 mmHg or DBP reading ≥110 mmHg within the 3 months before Day 1 or on Day 1).

18. Severe orthostatic hypotension despite optimal medical management (defined as a score of ≥3 on UMSARS Part I, Question 9).

Oncology 19. History of, or ongoing, malignant disease, including solid tumors and hematologic malignancies (with the exception of basal cell carcinomas and squamous cell carcinomas that have been completely excised and considered cured at least 12 months prior to Day -1). Participants with cancers in remission for greater than 5 years prior to Day -1 may be included.

Metabolic 20. Poorly controlled diabetes mellitus, as defined by having dosage adjustment of diabetic medication within 3 months before dosing (Day 1) or glycated hemoglobin value ≥8% at Baseline.

Hypersensitivity 21. Clinically significant allergies, as determined by the Investigator, to anesthetics that will be used for the LP per institutional practice, or iodine.

Other Medical History or Health Status 22. History of any clinically significant endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, renal ischemic, or other major diseases, as determined by the Investigator.

23. Surgery within 12 weeks before Day 1 (other than minor cosmetic surgery and minor dental surgery, as determined by the Investigator).

Any contraindications to LP procedures, including but not limited to:

24. Known or suspected structural abnormality of the lumbar spine, including but not limited to X-ray, MRI, or myelographic evidence of significant lumbar spine abnormalities, or other anatomical factors at or near the LP site that, in the opinion of the Investigator, may interfere with the performance of the LP, render repeated LPs difficult, or increase the risk of the procedure for the participant.

25. Presence of risk for increased or uncontrolled bleeding and/or risk of bleeding that is not managed optimally and might place a participant at an increased risk for intraoperative or postoperative bleeding. These could include, but are not limited to, anatomical factors at or near the LP site (e.g., vascular abnormalities, neoplasms, or other abnormalities), known underlying disorders of the coagulation cascade, platelet function, or platelet count (e.g., hemophilia, von Willebrand's disease, liver disease).

26. Unwillingness or inability to comply with the requirements of this protocol.

27. Other unspecified reasons that, in the opinion of the Investigator, make the participant unsuitable for enrollment.

Ages: 40 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Multiple system atrophy
Sampling Method: Non-Probability Sample
Enrollment: 29 (Actual)
Dates: Start 2020-06-17 (Actual); Primary Completion 2024-06-19 (Actual); Study Completion 2024-06-19 (Actual)

PRIMARY OUTCOMES:
Brain MRI imaging data | 5 years
  Diffusion-based MRI data
neurofilament light chain (NfL) in serum and/or plasma | 5 years
  Blood samples for measure measurement of NfL
Cerebral spinal fluid (CSF) measures | 5 years
  measurement of alpha synuclein, aggregated alpha synuclein Tau/phosphorylated Tau, neurofilament light chain, neurofilament heavy chain, and catecholamines in CSF
Quantitative movement assessment | 5 years
  The quantitative movement assessment comprises a battery of tests performed with non-invasive motion sensors, to capture disease features associated with striatonigral degeneration; others are aimed at capturing features associated with olivopontocerebellar degeneration observed in MSA patients.

CONTACTS AND LOCATIONS:
Overall Officials: Jose-Alberto Palma, MD PhD, Principal Investigator — NYU School of Medicine
Locations (1):
- NYU Langone Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Only de-identified, coded data will be shared with other researchers